CLINICAL TRIAL: NCT01903577
Title: Comparative Ergonomic Analysis of Robotic Versus Laparoscopic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Intuitive Surgical (Industry); Society of American Gastrointestinal and Endoscopic Surgeons (Other); Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Robotic Ergonomics-201101766
Record Dates: First submitted 2013-07-02; First posted 2013-07-19 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Ergonomics
Keywords: Ergonomics; Robotic Surgery; Laparoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Novice Laparoscopic and Robotic Surgeons (Experimental): Students and surgical trainees with less than 100 laparoscopic and less than 50 robotic cases.
  Will participate in Robotic Task Performance and Laparoscopic Task Performance
  Interventions: Other: Robotic Task Performance; Other: Laparoscopic Task Performance
- Expert Laparoscopists, Novice Roboticists (Experimental): Surgeons with more than 100 laparoscopic cases, less than 50 robotic cases.
  Will participate in Robotic Task Performance and Laparoscopic Task Performance
  Interventions: Other: Robotic Task Performance; Other: Laparoscopic Task Performance
- Expert robotic and laparoscopic surgeons (Experimental): Surgeons with greater than 100 laparoscopic and greater than 50 robotic cases.
  Will participate in Robotic Task Performance and Laparoscopic Task Performance
  Interventions: Other: Robotic Task Performance; Other: Laparoscopic Task Performance

INTERVENTIONS:
Other: Robotic Task Performance — Subjects will perform FLS tasks on the robotic platform while EMG data is being collected. Task performance and NASA task load index will be assessed. Experts in robotic surgery will also perform operative cases while EMG is being collected.
Other: Laparoscopic Task Performance — Subjects will perform FLS tasks on the laparoscopic platform while EMG data is being collected. Task performance and NASA task load index will be assessed. Experts in laparoscopic surgery will also perform operative cases while EMG is being collected.

SUMMARY:
Robotic surgery holds the potential to overcome many of the ergonomic challenges posed by laparoscopic surgery. In this study, we propose to quantify this potential ergonomic benefit by measuring electromyography (EMG) and instrument motion analysis of subjects performing surgical tasks using robotic assistance versus standard laparoscopic instrumentation.

Hypothesis: We hypothesize that surgeons will experience significant, measurable ergonomic advantages when performing tasks using robotic surgery when compared to conventional laparoscopic tools.

Study design: Subjects for the study will include three groups of varying degrees of training - (1) novice laparoscopists/novice roboticists, (2) expert laparoscopists/novice roboticists, and (3) expert laparoscopsts/expert roboticists. Subjects will perform the following tasks (chosen based on their reliability and validity in previous studies). Each task will be performed with standard laparoscopic instrumentation and with the da Vinci Surgical System.

* Inanimate (dry lab): Fundamentals of Laparoscopic (FLS) peg transfer, pattern cutting, intracorporeal suturing.
* Animate (porcine lab): laparoscopic bowel resection and anastomosis, robotic bowel resection and anastomosis.
* Human (clinical case): any laparoscopic or robotic procedure (preferably laparoscopic bowel resection and anastomosis, robotic bowel resection and anastomosis).

Outcome measures:

* Time to completion of tasks
* EMG: peak amplitudes, % maximum voluntary contraction and frequency analysis
* NASA Task Load Index scores
* Subject-Reported Qualitative Data from surveys
* Quality analysis of tasks (e.g., pattern cutting accuracy, % knots tied securely) for dry lab and animate lab tasks only)
* Instrument motion analysis of tasks (for dry lab and animate lab tasks only)

DETAILED DESCRIPTION:
Under an IRB-approved protocol, medical students, residents, fellows, and attending surgeons of the Department of Surgery and the Department of Obstetrics-Gynecology of Washington University School of Medicine who respond to the email or mailed letter invitation for recruitment will be screened by the Principal Investigator or one of the approved study members listed on the IRB protocol for inclusion and exclusion criteria using the following 5 screening questions:

1. What is your date of birth?
2. Are you a medical student, a resident, a fellow, or an attending surgeon in general surgery, urology, or obstetrics-gynecology?
3. Approximately how many laparoscopic surgeries have you performed as primary surgeon or first assistant surgeon during your career?
4. Approximately how many robotic surgeries have you performed as primary surgeon or first assistant surgeon during your career?
5. Do you have any known severe skin sensitivities or allergies to adhesives?

Those subjects who meet the inclusion criteria yet who are not disqualified by the exclusion criteria will be prospectively enrolled by an informed consent process into one of the three experimental groups of the study, defined by the subject's degrees of expertise in Minimally Invasive Surgery:

Inclusion Criteria:

1. age> 18 years
2. medical student, resident, fellow, or attending in Surgery, Urology, or Obstetrics-Gynecology at Washington University School of Medicine
3. Inclusion in Novice Laparoscopist/Novice Roboticist Group: performance of <100 laparoscopic cases and <50 robotic cases as primary surgeon or first assistant surgeon during one's career
4. Inclusion in Expert Laparoscopist/Novice Roboticist Group: performance of = or >100 laparoscopic cases and <50 robotic cases as primary surgeon or first assistant surgeon during one's career
5. Inclusion in Expert Laparoscopist/Expert Roboticist Group: performance of = or >100 laparoscopic cases and = or >50 robotic cases as primary surgeon or first assistant surgeon during one's career

Exclusion Criteria:

1. age <18 years
2. known severe skin sensitivities or allergies to adhesives

Screening, recruitment, and informed consent processes may be conducted by the Principal Investigator or any of the approved study members listed on the IRB protocol. To eliminate any potential for conflict of interest, recruitment and consent of medical students and residents for this study will be performed by a study investigator who does not have a supervisory role to medical students and residents, and not the Principal Investigator. To ensure that each subject is adequately informed of the study, the informed consent process will include but not be limited to discussion of the research procedures; anticipated frequency and types of participant interactions; length of the study period; potential risks and benefits to the participant; practices to protect the privacy and confidentiality of participants; the alternative to not participate in the clinical study; and means by which to ask questions, report concerns, or withdraw from the study at any time. Each subject will be informed that his decision to participate or not participate in the study does not in any way impact the health care decisions of his health care providers, or the clinical or academic performance evaluations of his evaluators. This information will also be included in the "Informed Consent Document" and the "Notice of Privacy Practices", and the content of these documents will be reviewed with each subject at the time of the informed consent discussion. Each subject will have the opportunity to review these documents at his leisure both before and after his decision to participate in the study, and each subject will receive at the time of the informed consent discussion a signed copy of the "Informed Consent Document" and the "Notice of Privacy Practices" to keep for his personal records. Each subject will be enrolled by informed consent discussion in a private environment to facilitate subject comfort in discussing details of the study and asking questions. During each subject enrollment attempt, the opportunity will be provided for the subject to meet individually with the approved study member listed on the IRB protocol to address private questions or concerns. Private environments may include a private office, a private conference room, or a private laboratory room. The subject will be able to discuss the study with family, friends, and/or others before deciding on participation. The subject will have until the end of the study enrollment period to consider study participation. Each subject who does not respond to the invitation to participate in the study at the time of the informed consent discussion will receive a copy of the "Informed Consent Document" and the "Notice of Privacy Practices" signed by the approved study member listed on the IRB protocol with whom informed consent was discussed, and a stamped envelope addressed to the Principal Investigator in the event that the subject wishes to consent to the study at a later time within the enrollment period. There will not be any follow-up contact regarding the study with subjects who do not wish to respond to the invitation to participate in the study. Capacity to consent for all subjects to be enrolled in the study will be determined by the approved study member listed on the IRB protocol conducting the informed consent. Capacity to consent will be assessed in a variety of ways such as explaining the study to the subject and then asking him to answer basic questions about the study procedures, risks and benefits, options for skipping questions, or how to withdraw from the study. The document entitled "Evaluation to Sign an Informed Consent" provided by the IRB may be a resource used to assist with this assessment. If at any time the approved study member listed on the IRB protocol has reason to believe that the subject is incompetent or incapacitated to make decisions for himself, the consent process will be aborted, and the subject will not be enrolled in the study.

ELIGIBILITY:
A) Novices Laparoscopists/Novice Roboticists

Inclusion Criteria:

1. age> 18 years
2. medical student, resident, fellow, or attending in Surgery, Urology, or Obstetrics-Gynecology at Washington University School of Medicine
3. performance of <100 laparoscopic cases and <50 robotic cases during one's career as primary surgeon or first assistant surgeon

Exclusion Criteria:

1. age <18 years
2. known severe skin sensitivities or allergies to adhesives

B) Expert Laparoscopists/Novice Roboticists

Inclusion Criteria:

1. age> 18 years
2. resident, fellow, or attending in Surgery, Urology, or Obstetrics-Gynecology at Washington University School of Medicine
3. performance of = or >100 laparoscopic cases during one's career and <50 robotic cases during one's career as primary surgeon or first assistant surgeon

Exclusion Criteria:

1. age <18 years
2. known severe skin sensitivities or allergies to adhesives

C) Expert Laparoscopists/Expert Roboticists

Inclusion Criteria:

1. age> 18 years
2. resident, fellow, or attending in Surgery, Urology, or Obstetrics-Gynecology at Washington University School of Medicine
3. performance of = or >100 laparoscopic cases and = or >50 robotic cases during one's career as primary surgeon or first assistant surgeon

Exclusion Criteria:

1. age <18 years
2. known severe skin sensitivities or allergies to adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
%MVC | At the time of Robotic and Laparoscopic Task Performance
  EMG: % maximum voluntary contraction will be calculated during each task repetition and surgical task

SECONDARY OUTCOMES:
Completion time | At the time of Robotic and Laparoscopic Task Performance
  Time to completion of tasks
NASA Task Load Index | At the time of Robotic and Laparoscopic Task Performance
  NASA Task Load Index scores in each of the six domains tested will be compared for laparoscopic and robotic surgical platforms
Quality analysis of tasks | At the time of Robotic and Laparoscopic Task Performance
  Quality analysis of tasks performed (pattern cutting accuracy, % knots tied securely) for dry lab tasks only

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Awad, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St Louis School of Medicine, St Louis, Missouri, United States